CLINICAL TRIAL: NCT02431338
Title: Cost-effectiveness of Remote Ischemic Conditioning as an Adjunct to Primary Percutaneous Coronary Intervention in Patients With ST-elevation Myocardial Infarction
Brief Title: Cost-effectiveness of Remote Ischemic Conditioning as an Adjunct to Primary Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48241
Record Dates: First submitted 2015-04-17; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: Remote ischemic conditioning; Cost-effectiveness analysis
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Remote ischemic conditioning through intermittent arm ischemia with four cycles of alternating 5-minute inflation followed by 5-minute deflation of a blood pressure cuff performed in the ambulance during transport to primary percutaneous coronary intervention.
  Interventions: Procedure: Remote ischemic conditioning
- Control group (No Intervention): Standard treatment with primary percutaneous coronary intervention alone.

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Intermittent arm ischemia through four cycles of alternating 5-minute inflation followed by 5-minute deflation of a blood pressure cuff placed around the upper arm.
  Other Names: RIC
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate the cost-effectiveness of remote ischemic conditioning as an adjunct to primary percutaneous coronary intervention from the perspective of a Danish healthcare system.

ELIGIBILITY:
Inclusion Criteria:

(1) age ≥ 18 years, (2) symptom duration of ≤ 12 hours prior to admission, and (3) ST-segment elevation ≥ 0.1 mV in two or more contiguous electrocardiogram (ECG) leads

Exclusion Criteria:

(1) diagnosis not confirmed during hospital admission, (2) history of previous myocardial infarction, (3) previous CABG, and (4) chest pain > 12 hours prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2007-02; Primary Completion 2012-01 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Incremental cost-effectiveness ratio (ICER) = [difference in total cardiovascular medical care costs between treatment groups] / [difference in major adverse cardiac and cerebrovascular event (MACCE)-free survival between treatment groups] | 4-years of follow-up
  Data for the economic evaluation are collected from Danish nationwide registries and validated with medical record review. Charges from the Diagnosis Related Group (DRG) and the Danish Ambulatory Grouping System /DAGS) are used to calculate total cardiovascular medical care costs in the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid D Sloth, MD, Principal Investigator — Department of Cardiology, Aarhus University Hospital, Denmark
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Aarhus N, Denmark